CLINICAL TRIAL: NCT01850446
Title: Comparative Parallel-group Randomized Clinical Trial of Efficacy and Safety of Ergoferon Versus Oseltamivir in Treatment of Influenza
Brief Title: Comparative Clinical Trial of Efficacy and Safety of Ergoferon Versus Oseltamivir in Treatment of Influenza
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMH-ER-003
Record Dates: First submitted 2013-04-30; First posted 2013-05-09 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2019-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — ergoferon; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergoferon (Experimental): The treatment period is 5 days. Oral Dose per administration: 1 tablet. The tablet should be kept in the mouth until completely dissolution, the drug is taken without regard to food intake.
  Interventions: Drug: Ergoferon
- Oseltamivir (Tamiflu) (Active Comparator): The treatment period is 5 days.
  1 capsule (75 mg) twice a day during the meal or regardless of meal.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Ergoferon — Safety and Efficacy
  Arms: Ergoferon
Drug: Oseltamivir — Safety and Efficacy
  Other Names: Tamiflu
  Arms: Oseltamivir (Tamiflu)

SUMMARY:
The purpose of this study is:

* to assess the efficacy of Ergoferon in treatment of influenza;
* to assess the safety of Ergoferon in treatment of influenza;
* to compare the efficacy of Ergoferon and Oseltamivir for treatment of influenza.

DETAILED DESCRIPTION:
The overall duration of a patient participation in the trial is 6 days (screening/randomization/therapy onset - day 1; study therapy period - day 1-5; follow-up period - day 6).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70 years.
2. Patients who were admitted to hospital within 48 hours from the onset of influenza signs.
3. Patients with body temperature ≥37,8°C when visiting a doctor + severity of influenza symptoms ≥4 scores (presence of at least 1 non-specific flu symptom ≥2 scores and 1 nasal/ throat/ chest symptom ≥ 2 scores or greater number of symptoms with the severity ≥1 score).
4. Diagnosed influenza confirmed by rapid diagnostic test (OSOM Influenza A&B Test).
5. The possibility to start therapy within 48 hours after the onset of the first symptoms of influenza.
6. Usage of contraceptive methods by both gender patients of reproductive age during the trial and within 30 days after ending the participation in the trial.
7. Availability of signed patient information sheet (Informed Consent form) for participation in the clinical trial.

Exclusion Criteria:

1. Suspected pneumonia, bacterial infection or the presence of a severe disease requiring usage of antibacterial drugs (including sulphanilamides) starting from Day 1 of the disease.
2. Severe influenza with indications for hospitalization.
3. Suspected early manifestations of diseases that have symptoms similar to influenza symptoms (other acute respiratory and infectious diseases, influenza-like syndrome at the onset of systemic connective tissue disorders, hematologic neoplasms and other pathology).
4. Patients requiring concurrent antiviral products forbidden by the study.
5. Medical history of primary and secondary immunodeficiencies. а) lymphoid immunodeficiencies (Т-cell and/or В-cell, immunodeficiencies with predominant antibody deficit); b) phagocytic deficits; c) complement factor deficit; d) combined immunodeficiencies including AIDS secondary to HIV infection; toxic, autoimmune, infectious, radiation panleukopenic syndrome; total lymphocytopenic syndrome; polyclonal lymphocyte activation syndrome; postsplenectomic syndrome; congenital asplenia; abnormal immune complex syndrome associated with infectious, autoimmune and allergic diseases.
6. Medical history of sarcoidosis
7. An oncological disease/suspected oncological disease.
8. Exacerbated or decompensated chronic diseases affecting a patient's ability to participate in the clinical trial.
9. Medical history of polyvalent allergy.
10. Allergy/intolerance to any of the components of the product used for influenza therapy.
11. Impaired glucose tolerance, type 1 and type 2 diabetes mellitus.
12. Malabsorption syndrome, including congenital or acquired lactose deficiency or another disaccharide deficiency.
13. Pregnancy, breast-feeding.
14. Consumption of narcotics, alcohol > 2 alcohol units per day, mental diseases.
15. Use of any medicine listed in the section "Prohibited concomitant treatment" within 30 days preceding the inclusion in this study.
16. Patients who, from the investigator's point of view, will fail to comply with the observation requirements of the trial or with the regimen of the study drugs.
17. Participation in other clinical studies within 1 month prior to enrollment in the current trial.
18. Patients related to the research staff of the clinical trial site who are directly involved in the trial or are the immediate family member of the researcher. The immediate family members include husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
19. Patients employed with OOO "NPF "MATERIA MEDICA HOLDING" (i.e., the company's employee, part-time employee under contract, or appointed official in charge of the trial, or their immediate family).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - The Non-State Health Care Institution "Road Hospital of the Open Joint Stock Company" Russian Railways", Chelyabinsk
  - The State Budgetary Educational Institution of Higher Professional Education " Kazan State University of Medicine" Ministry of Health of the Russian Federation, Kazan'
  - Pirogov Russian National Research Medical University, Moscow
  - Federal State Budgetary Military Educational Institution of Higher Professional Education "Military-Medicine Academy named after S. M. Kirov" of Ministry of Defence of Russian Federation, Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution " City policlinic No. 117", Saint Petersburg
  - Limited Liability Company "Scientific Research Centre Eco-safety", Saint Petersburg
  - Regional State Budgetary Healthcare Institution "Clinical Hospital №1", Smolensk

RESULTS

PARTICIPANT FLOW:
Groups:
- Ergoferon (1 Tablet 3 Times a Day): Ergoferon: The treatment period is 5 days. Oral Dose per administration: 1 tablet. The tablet should be kept in the mouth until completely dissolution, the drug is taken without regard to food intake.
  Dosing scheme. One tablet every 30 minutes for the first 2 hours, then during the first day, three more doses are taken at equal intervals. From the second to the fifth day, the drug is taken 1 tablet 3 times a day.
- Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day: Oseltamivir: The treatment period is 5 days.
  1 capsule (75 mg) twice a day during the meal or regardless of meal.
Period: Overall Study
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Started | 92 | 92
Completed | 87 | 90
Not Completed | 5 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (13.7) | 38.4 (14.4) | 38.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 46 | 99
  Male | 39 | 46 | 85
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Count of Participants [Count of Participants; unit: Participants] | 92 | 92 | 184

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Recovery/Improvement in Health Status.
Description: Based on days 2-7 days of observation according to the patient's diary, and on days 3 and 7 according to the physician's examination.
Time Frame: On 2-7 days of observation
Population: Intention to treat [ITT]
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
Participants
  Morning, day 2 (patient diary data) | 2 | 3
  Morning, day 3 (patient diary data) | 2 | 3
  Morning, day 4 (patient diary data) | 7 | 9
  Morning, day 5 (patient diary data) | 31 | 21
  Morning, day 6 (patient diary data) | 49 | 49
  Morning, day 7 (patient diary data) | 68 | 62
  Evening, day 2 (patient diary data) | 1 | 4
  Evening, day 3 (patient diary data) | 3 | 6
  Evening, day 4 (patient diary data) | 12 | 9
  Evening, day 5 (patient diary data) | 36 | 31
  Evening, day 6 (patient diary data) | 60 | 53
  Day 3 (physician's examination): number analyzed (Participants) | 87 | 92
  Day 3 (physician's examination) | 2 | 5
  Day 7 (physician's examination): number analyzed (Participants) | 87 | 92
  Day 7 (physician's examination) | 69 | 68
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Individual day analyses were combined into Global Test Statistics (patient diary analysis); Test type: Non-Inferiority — Non-inferiority margin was prespecified as 20% (on each day). Type I error (alpha) level of 0.025 was prospectively planned for this analysis. Power of this analysis was planned to be greater than 0.8; p < 0.0001, Z-test for Global test statistics — Global test statistics (GTS) was constructed in accordance with O'Brien Procedures for Comparing Samples with Multiple Endpoints; Z-value = 8.56
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Individual day analyses were combined into Global Test Statistics (physician's examination analysis); Test type: Non-Inferiority — Non-inferiority margin was prespecified as 20% (on each day). Type I error (alpha) level of 0.025 was prospectievely planned for this analysis. Power of this analysis was planned to be greater than 0.8; p < 0.0001, Z-test for Global test statistics — Global test statistics (GTS) was constructed in accordance with O'Brien, P. (1984). Procedures for Comparing Samples with Multiple Endpoints. Biometrics, 40(4), 1079-1087. doi:10.2307/2531158; Z-value = 7.31

2. Secondary Outcome: Changes in Fever.
Description: Fever changes over time (body temperature change on days 2-7 compared to baseline, based on patient diary data).
Time Frame: Baseline and days 2-7 of the observation
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
°C
  Morning, day 1 | 38.8 (0.5) | 38.7 (0.5)
  Morning, day 2 | 37.8 (0.7) | 37.8 (0.8)
  Morning, day 3 | 37.4 (0.6) | 37.2 (0.7)
  Morning, day 4 | 37.0 (0.5) | 36.9 (0.5)
  Morning, day 5 | 36.8 (0.4) | 36.7 (0.5)
  Morning, day 6 | 36.6 (0.3) | 36.6 (0.4)
  Morning, day 7 | 36.5 (0.3) | 36.5 (0.3)
  Evening, day 1 | 38.3 (0.7) | 38.3 (0.8)
  Evening, day 2 | 37.8 (0.6) | 37.7 (0.8)
  Evening, day 3 | 37.3 (0.5) | 37.2 (0.7)
  Evening, day 4 | 37.0 (0.4) | 37.0 (0.5)
  Evening, day 5 | 36.8 (0.4) | 36.8 (0.4)
  Evening, day 6 | 36.6 (0.3) | 36.7 (0.4)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of fever was measured as area under curve (body temperature-time); Test type: Non-Inferiority — Non-inferiority margin was prespecified as 1.2 degree*day; p = 0.027, t-test, 1 sided; Mean Difference (Final Values) = 0.44, 97.5% CI 1-sided [lower limit -0.23]

3. Secondary Outcome: Average Duration of Fever.
Description: Criteria of no fever - body temperature lower than 37.0° C for 24 hours
Time Frame: From the time of randomization until the time of recovery/improvement (days 1-7)
Population: Intention to treat (ITT)
Measure: Mean (Standard Error); unit: days
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
days | 3.77 (0.13) | 3.54 (0.16)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Test type: Non-Inferiority — Non-inferiority magrin was prespecified as 20% of comparator duration; p = 0.02, t-test, 1 sided; mean survival time estimates obtained from survival analysis were compared by means of t-test with infinite degrees of freedom; Mean Difference (Final Values) = 0.23, 97.5% CI 1-sided [upper limit 0.63]

4. Secondary Outcome: Percentage of Patients With Normal Body Temperature.
Description: Based on patient's diary. Normal body temperature is no more than 37.0ºС.
Time Frame: Days 2-7 of the observation
Population: Intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
Participants
  Morning, day 2 | 11 | 12
  Morning, day 3 | 21 | 31
  Morning, day 4 | 43 | 49
  Morning, day 5 | 68 | 72
  Morning, day 6 | 83 | 81
  Morning, day 7 | 90 | 88
  Evening, day 2 | 9 | 20
  Evening, day 3 | 17 | 29
  Evening, day 4 | 45 | 48
  Evening, day 5 | 69 | 69
  Evening, day 6 | 83 | 78
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Individual day analyses were combined into Global Test Statistics; Test type: Non-Inferiority — Non-inferiority margin was prespecified as 20% (on each day); p < 0.0001, Z-test for Global test statistics — [p-value comment as in outcome 1, analysis 2]; Z-value = 6.95

5. Secondary Outcome: Severity of Influenza Symptoms (Fever, Flu Non-specific and Nasal/Throat/Chest Symptoms) in Scores According to the Symptoms Severity Scale.
Description: The symptoms severity scale includes 14 symptoms: body temperature, non-specific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness), nasal/throat/chest symptoms (runny nose, stuffy nose, sneezing, sore throat, hoarseness, cough, chest pain).
  The severity of each non-specific and nasal/throat/chest symptom is scored on a 4-point scale (0=no symptom; 1=mild symptom; 2=moderate symptom; 3=severe symptom). The minimum value of each symptom is 0 points, and the maximum value is 4 points.
  The absolute body temperature (in degrees Celsius) is converted to relative units (or scores) using the following scale: ≤37.2С=0 points; 37.3-38.0С=1 point; 38.1-39.0С=2 points; ≥39.1С=3 points.
  The severity of symptoms is based on the physical examination of the patient by the physician on days 1, 3, and 7 and on the patient diary data on days 1-7. The minimum symptoms severity score is 0 points, the maximum score is 42 points.
Time Frame: On 1-7 days of observation
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
score on a scale
  Morning, day 1 (patient diary data) | 20.4 (6.5) | 20.9 (5.9)
  Morning, day 2 (patient diary data) | 16.3 (6.8) | 15.7 (7.1)
  Morning, day 3 (patient diary data) | 13.0 (6.6) | 12.2 (5.9)
  Morning, day 4 (patient diary data) | 8.7 (5.3) | 8.0 (5.4)
  Morning, day 5 (patient diary data) | 5.4 (4.8) | 5.7 (4.3)
  Morning, day 6 (patient diary data) | 3.6 (3.7) | 3.7 (3.4)
  Morning, day 7 (patient diary data) | 2.3 (3.5) | 2.5 (3.1)
  Evening, day 1 (patient diary data) | 18.8 (6.8) | 18.2 (7.0)
  Evening, day 2 (patient diary data) | 15.6 (7.0) | 14.7 (6.9)
  Evening, day 3 (patient diary data) | 11.4 (6.1) | 10.1 (5.7)
  Evening, day 4 (patient diary data) | 7.2 (5.0) | 7.3 (4.9)
  Evening, day 5 (patient diary data) | 4.9 (4.4) | 4.6 (4.0)
  Evening, day 6 (patient diary data) | 2.9 (3.6) | 3.2 (3.4)
  Day 1 (based on physician's objective examination) | 19.7 (6.6) | 20.1 (6.1)
  Day 3 (based on physician's objective examination) | 12.7 (6.3) | 11.3 (5.7)
  Day 7 (based on physician's objective examination) | 2.0 (3.1) | 2.0 (2.5)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day1 morning); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -0.49, 97.5% CI 1-sided [upper limit 1.33]
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day2 morning); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.013, t-test, 1 sided; Mean Difference (Final Values) = 0.56, 97.5% CI 1-sided [upper limit 2.59]
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day3 morning); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.084, t-test, 1 sided; Mean Difference (Final Values) = 0.82, 97.5% CI 1-sided [upper limit 2.66]
Statistical Analysis 4: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day4 morning); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.22, t-test, 1 sided; Mean Difference (Final Values) = 0.62, 97.5% CI 1-sided [upper limit 2.2]
Statistical Analysis 5: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day5 morning); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.04, t-test, 1 sided; Mean Difference (Final Values) = -0.27, 97.5% CI 1-sided [upper limit 1.07]
Statistical Analysis 6: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day6 morning); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.13, t-test, 1 sided; Mean Difference (Final Values) = -0.08, 97.5% CI 1-sided [upper limit 0.98]
Statistical Analysis 7: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; severity of influenza symptoms (day1 morning); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.135, t-test, 1 sided; Mean Difference (Final Values) = -0.25, 97.5% CI 1-sided [upper limit 0.74]
Statistical Analysis 8: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day1 evening); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.004, t-test, 1 sided; Mean Difference (Final Values) = 0.64, 97.5% CI 1-sided [upper limit 2.67]
Statistical Analysis 9: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day2 evening); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.05, t-test, 1 sided; Mean Difference (Final Values) = 0.9, 97.5% CI 1-sided [upper limit 2.94]
Statistical Analysis 10: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day3 evening); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.447, t-test, 1 sided; Mean Difference (Final Values) = 1.34, 97.5% CI 1-sided [upper limit 3.08]
Statistical Analysis 11: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day4 evening); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.042, t-test, 1 sided; Mean Difference (Final Values) = -0.08, 97.5% CI 1-sided [upper limit 1.4]
Statistical Analysis 12: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day5 evening); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.313, t-test, 1 sided; Mean Difference (Final Values) = 0.29, 97.5% CI 1-sided [upper limit 1.53]
Statistical Analysis 13: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day6 evening); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.087, t-test, 1 sided; Mean Difference (Final Values) = -0.27, 97.5% CI 1-sided [upper limit 0.77]
Statistical Analysis 14: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day1 physician's objective examination); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -0.43, 97.5% CI 1-sided [upper limit 1.41]
Statistical Analysis 15: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza symptoms (day3 physician's objective examination); Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.305, t-test, 1 sided; Mean Difference (Final Values) = 1.34, 97.5% CI 1-sided [upper limit 3.11]

6. Secondary Outcome: Duration of Clinical Symptoms of Influenza (Fever, Non-specific Symptoms and Nasal/ Throat/ Chest Symptoms) in Days.
Description: Duration of clinical symptoms of influenza (fever, non-specific symptoms and nasal/ throat/ chest symptoms) in days based on the result of the patient's diary data
Time Frame: On 1-7 days of observation
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
days
  Fever | 2.96 (0.13) | 2.86 (0.16)
  Non-specific symptoms | 4.82 (0.12) | 5.0 (0.11)
  Nasal/ throat/ chest symptoms | 4.83 (0.15) | 5.08 (0.11)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Fever duration; Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p = 0.02, t-test, 1 sided; Mean Difference (Final Values) = 0.08, 97.5% CI 1-sided [upper limit 0.5]
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Non-specific symptoms duration; Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -0.18, 97.5% CI 1-sided [upper limit 0.14]
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Nasal/ throat/ chest symptoms duration; Test type: Non-Inferiority — N.I. margin was prespecified as 20% of comparator (with respect to timeframe); p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = -0.25, 97.5% CI 1-sided [upper limit 0.11]

7. Secondary Outcome: The Severity of Influenza.
Description: Based on the patient diary. The severity of influenza based on the data on the "Area Under Curve" for total index of influenza severity.
Time Frame: On days 1-7 of the observation.
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score*day
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
score*day | 59.88 (24.82) | 57.88 (25.08)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Severity of influenza was measured as area under curve (symptoms score-time); Test type: Non-Inferiority — N.I. margin was prespecified as 20% (AUC ratio supposed to be less than 1.2); p = 0.015, one-sample Z-test — bootstrap (100000 rep) confidence limits were constructed for AUC ratio; AUC ratio was compared with N.I. margin; AUC ratio = 1.04, 95% CI 2-sided [0.9 to 1.17]

8. Secondary Outcome: Percentage of Patients Who Used Antipyretics on Days 1, 2, 3, 4 and 5 of the Treatment.
Description: Antipyretics, which are allowed for use during clinical trial, are:
  1. Paracetamol;
  2. Metamizole sodium (if hyperthermia was not stopped by usage of paracetamol).
Time Frame: Days 1, 2, 3, 4 and 5 of the treatment
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
Participants
  Day 1 | 64 | 59
  Day 2 | 39 | 38
  Day 3 | 14 | 11
  Day 4 | 1 | 3
  Day 5 | 0 | 2
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Percentage difference of Patients, Who Used Antipyretics (day1); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p = 0.036, Z test for proportions; Risk Difference (RD) = 0.05, 97.5% CI 1-sided [upper limit 0.19]
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Percentage difference of Patients, Who Used Antipyretics (day2); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p = 0.009, Z test for proportions; Risk Difference (RD) = 0.01, 97.5% CI 1-sided [upper limit 0.15]
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Percentage difference of Patients, Who Used Antipyretics (day3); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p < 0.001, Z test for proportions; Risk Difference (RD) = 0.03, 97.5% CI 1-sided [upper limit 0.13]
Statistical Analysis 4: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Percentage difference of Patients, Who Used Antipyretics (day4); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p < 0.001, Z test for proportions; Risk Difference (RD) = -0.02, 97.5% CI 1-sided [upper limit 0.13]
Statistical Analysis 5: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Percentage difference of Patients, Who Used Antipyretics (day5); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p < 0.001, Z test for proportions; Risk Difference (RD) = -0.02, 97.5% CI 1-sided [upper limit 0.01]

9. Secondary Outcome: Percentage of Patients Requiring Antibiotics Administration.
Description: Based on patient's diary, objective examination (according to physician's objective examination).
  The patients with the development of disease complications and exacerbation of the disease course (the development of severe influenza).
Time Frame: On 1-7 days of observation.
Population: Intention to treat [ITT]
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 92 | 92
Participants | 1 | 1
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Percentage of Patients Requiring Antibiotics Administration; Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p < 0.001, Z test for proportions; Risk Difference (RD) = 0, 97.5% CI 1-sided [upper limit 0.03]

10. Secondary Outcome: Proportion of Patients With Negative Results of Virological Analysis.
Description: Based on medical records of patients whose nasopharyngeal swabs submitted for Reverse Transcription Polymerase Chain Reaction (RT-PCR) were negative for influenza A/B virus.
Time Frame: On days 3, 5, 7 of observation.
Population: The number of patients to whom RT-PCR of the nasal samples was performed does not match the total number of patients in the ITT set due to the fact that not all nasopharyngeal samples were tested (due to violations of storage conditions in the centres before their transportation to the central laboratory).
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 69 | 77
Participants
  Day 3 | 45 | 50
  Day 5 | 57 | 70
  Day 7 | 65 | 75
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Proportion difference of Patients With Negative Results (day3); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p = 0.014, Z test for proportions; Risk Difference (RD) = -0.01, 97.5% CI 1-sided [upper limit 0.15]
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Proportion difference of Patients With Negative Results (day5); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p = 0.037, Z test for proportions; Risk Difference (RD) = -0.08, 97.5% CI 1-sided [upper limit 0.03]
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; Proportion difference of Patients With Negative Results (day7); Test type: Non-Inferiority — N.I. margin was prespecified as 20%; p < 0.001, Z test for proportions; Risk Difference (RD) = -0.03, 97.5% CI 1-sided [upper limit 0.03]

11. Secondary Outcome: Dynamics of Parameters of Immune Status (T-cell and B-cell Immune Response).
Description: The concentration of regulators of the T-cell immune response (IL2, IFN -γ, IL-18), and regulators of В-cell immune response (IL-4, IL-16).
Time Frame: On days1, 3 and 7 of observation.
Population: Intention to treat [ITT]
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 19 | 31
pg/mL
  IL-2/Day1 | 3.25 (2.70) | 4.26 (3.38)
  IL-2/Day3 | 4.40 (4.31) | 3.52 (2.59)
  IL-2/Day7: number analyzed (Participants) | 18 | 30
  IL-2/Day7 | 4.65 (4.07) | 4.39 (3.29)
  IFN-γ/Day1 | 5.11 (2.28) | 9.91 (8.78)
  IFN-γ/Day3 | 7.21 (4.24) | 7.76 (5.25)
  IFN-γ/Day7: number analyzed (Participants) | 18 | 30
  IFN-γ/Day7 | 9.00 (5.25) | 6.63 (11.03)
  IL-18/Day1 | 238.99 (138.86) | 192.15 (119.85)
  IL-18/Day3 | 277.74 (188.73) | 220.64 (152.33)
  IL-18/Day7: number analyzed (Participants) | 18 | 30
  IL-18/Day7 | 239.84 (140.24) | 195.01 (134.45)
  IL-4/Day1 | 1.26 (1.40) | 1.39 (0.75)
  IL-4/Day3 | 1.54 (1.83) | 1.21 (0.61)
  IL-4/Day7: number analyzed (Participants) | 18 | 30
  IL-4/Day7 | 1.51 (1.41) | 1.32 (0.55)
  IL-16/Day1 | 28.40 (30.16) | 60.41 (46.37)
  IL-16/Day3 | 44.26 (75.11) | 58.15 (46.15)
  IL-16/Day7: number analyzed (Participants) | 18 | 29
  IL-16/Day7 | 45.36 (74.18) | 64.45 (44.13)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (IL-2); Test type: Superiority; p = 0.03, t-test, 2 sided — P-value IL2 provided for between-group comparisson of difference from days 3 to day 1; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [0.19 to 3.59]
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (IL-2); Test type: Superiority; p = 0.19, t-test, 2 sided — P-value IL2 provided for between-group comparisson of difference from day 7 to day 1; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-0.64 to 3.12]
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (IFN-γ); Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (IFN-γ); Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (IL-18); Test type: Superiority; p = 0.795, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (IL-18); Test type: Superiority; p = 0.992, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (IL-4); Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [0.02 to 0.92]
Statistical Analysis 8: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (IL-4); Test type: Superiority; p = 0.08, t-test, 2 sided; Median Difference (Final Values) = 0.37, 95% CI 2-sided [-0.04 to 0.79]
Statistical Analysis 9: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (IL-16); Test type: Superiority; p = 0.062, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (IL-16); Test type: Superiority; p = 0.638, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Dynamics of Parameters of Immune Status ( IFN-α and IFN-γ Production).
Description: Level of spontaneous and induced production of IFN-α and IFN-γ (in vitro).
Time Frame: On day 1, 3 and 7 of observation.
Population: Intention to treat [ITT]
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 19 | 31
pg/mL
  Spontaneous IFN-α/Day1: number analyzed (Participants) | 12 | 21
  Spontaneous IFN-α/Day1 | 11.42 (5.01) | 8.25 (7.91)
  Spontaneous IFN-α/Day3: number analyzed (Participants) | 11 | 21
  Spontaneous IFN-α/Day3 | 12.39 (6.20) | 6.19 (4.33)
  Spontaneous IFN-α/Day7: number analyzed (Participants) | 6 | 18
  Spontaneous IFN-α/Day7 | 8.04 (4.36) | 6.12 (4.00)
  Induced IFN-α/Day1: number analyzed (Participants) | 12 | 21
  Induced IFN-α/Day1 | 13.30 (5.52) | 13.58 (11.31)
  Induced IFN-α/Day3: number analyzed (Participants) | 11 | 21
  Induced IFN-α/Day3 | 12.98 (4.51) | 9.73 (6.48)
  Induced IFN-α/Day7: number analyzed (Participants) | 6 | 18
  Induced IFN-α/Day7 | 9.06 (2.22) | 8.55 (4.16)
  Spontaneous IFN-γ/Day1: number analyzed (Participants) | 12 | 21
  Spontaneous IFN-γ/Day1 | 14.27 (6.15) | 10.73 (7.33)
  Spontaneous IFN-γ/Day3: number analyzed (Participants) | 11 | 21
  Spontaneous IFN-γ/Day3 | 20.79 (21.16) | 11.99 (12.34)
  Spontaneous IFN-γ/Day7: number analyzed (Participants) | 6 | 19
  Spontaneous IFN-γ/Day7 | 10.34 (6.30) | 17.00 (23.99)
  Induced IFN-γ/Day1: number analyzed (Participants) | 12 | 21
  Induced IFN-γ/Day1 | 113.31 (157.45) | 164.92 (156.01)
  Induced IFN-γ/Day3: number analyzed (Participants) | 11 | 21
  Induced IFN-γ/Day3 | 84.16 (75.58) | 177.92 (208.27)
  Induced IFN-γ/Day7: number analyzed (Participants) | 6 | 18
  Induced IFN-γ/Day7 | 95.16 (82.51) | 154.31 (156.57)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (Spontaneous IFN-α); Test type: Superiority; p = 0.065, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (Spontaneous IFN-α); Test type: Superiority; p = 0.404, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (Induced IFN-α); Test type: Superiority; p = 0.204, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (Induced IFN-α); Test type: Superiority; p = 0.386, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (Spontaneous IFN-γ); Test type: Superiority; p = 0.592, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (Spontaneous IFN-γ); Test type: Superiority; p = 0.356, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (Induced IFN-γ); Test type: Superiority; p = 0.475, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (Induced IFN-γ); Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Dynamics of Parameters of Immune Status (Absolute Number of Each Type of White Blood Cells and Different Lymphocyte Phenotypes).
Description: The absolute number of each type of white blood cells (WBC): Absolut Count (AC) of leukocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils, and CD3, CD4, CD8, CD4/CD8, CD16, CD119 leukocytes.
Time Frame: On days 1, 3 and 7 of observation.
Population: Intention to treat [ITT]
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 19 | 31
10^9 cells/L
  AC of leukocytes/Day1: number analyzed (Participants) | 19 | 29
  AC of leukocytes/Day1 | 5.47 (1.74) | 5.33 (1.57)
  AC of leukocytes/Day3: number analyzed (Participants) | 18 | 31
  AC of leukocytes/Day3 | 4.98 (1.73) | 4.61 (1.49)
  AC of leukocytes/Day7: number analyzed (Participants) | 18 | 27
  AC of leukocytes/Day7 | 5.81 (1.96) | 6.50 (1.80)
  AC of neutrophils/Day1: number analyzed (Participants) | 19 | 29
  AC of neutrophils/Day1 | 3.39 (1.43) | 3.23 (1.25)
  AC of neutrophils/Day3: number analyzed (Participants) | 18 | 31
  AC of neutrophils/Day3 | 2.32 (1.08) | 2.13 (1.12)
  AC of neutrophils/Day7: number analyzed (Participants) | 18 | 27
  AC of neutrophils/Day7 | 2.73 (1.28) | 3.45 (1.54)
  AC of lymphocytes/Day1: number analyzed (Participants) | 19 | 29
  AC of lymphocytes/Day1 | 1.37 (0.67) | 1.26 (0.48)
  AC of lymphocytes/Day3: number analyzed (Participants) | 18 | 31
  AC of lymphocytes/Day3 | 1.98 (0.69) | 1.86 (0.57)
  AC of lymphocytes/Day7: number analyzed (Participants) | 18 | 27
  AC of lymphocytes/Day7 | 2.46 (0.91) | 2.41 (0.63)
  AC of monocytes/Day1: number analyzed (Participants) | 19 | 29
  AC of monocytes/Day1 | 0.62 (0.30) | 0.73 (0.27)
  AC of monocytes/Day3: number analyzed (Participants) | 18 | 31
  AC of monocytes/Day3 | 0.58 (0.25) | 0.50 (0.20)
  AC of monocytes/Day7: number analyzed (Participants) | 18 | 27
  AC of monocytes/Day7 | 0.47 (0.18) | 0.49 (0.21)
  AC of eosinophils/Day1: number analyzed (Participants) | 19 | 29
  AC of eosinophils/Day1 | 0.06 (0.06) | 0.07 (0.09)
  AC of eosinophils/Day3: number analyzed (Participants) | 18 | 31
  AC of eosinophils/Day3 | 0.07 (0.06) | 0.10 (0.09)
  AC of eosinophils/Day7: number analyzed (Participants) | 18 | 27
  AC of eosinophils/Day7 | 0.11 (0.09) | 0.12 (0.11)
  AC of basophils/Day1: number analyzed (Participants) | 19 | 29
  AC of basophils/Day1 | 0.03 (0.02) | 0.04 (0.04)
  AC of basophils/Day3: number analyzed (Participants) | 18 | 31
  AC of basophils/Day3 | 0.02 (0.02) | 0.03 (0.02)
  AC of basophils/Day7: number analyzed (Participants) | 18 | 27
  AC of basophils/Day7 | 0.04 (0.02) | 0.03 (0.02)
  AC of CD3+/Day1 | 1.06 (0.60) | 1.17 (0.91)
  AC of CD3+/Day3: number analyzed (Participants) | 19 | 30
  AC of CD3+/Day3 | 1.59 (0.55) | 1.48 (0.54)
  AC of CD3+/Day7: number analyzed (Participants) | 14 | 27
  AC of CD3+/Day7 | 1.89 (0.77) | 1.86 (0.57)
  AC of CD3+CD4+/Day1 | 0.66 (0.41) | 0.74 (0.61)
  AC of CD3+CD4+/Day3: number analyzed (Participants) | 19 | 30
  AC of CD3+CD4+/Day3 | 1.02 (0.39) | 0.95 (0.38)
  AC of CD3+CD4+/Day7: number analyzed (Participants) | 14 | 27
  AC of CD3+CD4+/Day7 | 1.24 (0.60) | 1.22 (0.46)
  AC of CD3+CD8+/Day1 | 0.36 (0.22) | 0.38 (0.33)
  AC of CD3+CD8+/Day3: number analyzed (Participants) | 19 | 30
  AC of CD3+CD8+/Day3 | 0.52 (0.22) | 0.47 (0.20)
  AC of CD3+CD8+/Day7: number analyzed (Participants) | 14 | 27
  AC of CD3+CD8+/Day7 | 0.61 (0.28) | 0.59 (0.19)
  AC of CD3+CD16+CD56+/Day1 | 0.07 (0.06) | 0.09 (0.16)
  AC of CD3+CD16+CD56+/Day3: number analyzed (Participants) | 19 | 30
  AC of CD3+CD16+CD56+/Day3 | 0.11 (0.09) | 0.07 (0.04)
  AC of CD3+CD16+CD56+/Day7: number analyzed (Participants) | 14 | 27
  AC of CD3+CD16+CD56+/Day7 | 0.10 (0.10) | 0.07 (0.05)
  AC of CD3-CD16+CD56+/Day1 | 0.15 (0.11) | 0.16 (0.18)
  AC of CD3-CD16+CD56+/Day3: number analyzed (Participants) | 19 | 30
  AC of CD3-CD16+CD56+/Day3 | 0.19 (0.14) | 0.16 (0.13)
  AC of CD3-CD16+CD56+/Day7: number analyzed (Participants) | 14 | 27
  AC of CD3-CD16+CD56+/Day7 | 0.17 (0.15) | 0.17 (0.11)
  AC of CD3-CD8+/Day1 | 0.05 (0.03) | 0.06 (0.09)
  AC of CD3-CD8+/Day3: number analyzed (Participants) | 19 | 30
  AC of CD3-CD8+/Day3 | 0.08 (0.06) | 0.07 (0.05)
  AC of CD3-CD8+/Day7: number analyzed (Participants) | 14 | 27
  AC of CD3-CD8+/Day7 | 0.09 (0.07) | 0.07 (0.05)
  AC of CD19+CD3-/Day1 | 0.19 (0.14) | 0.20 (0.12)
  AC of CD19+CD3-/Day3: number analyzed (Participants) | 19 | 30
  AC of CD19+CD3-/Day3 | 0.20 (0.15) | 0.20 (0.09)
  AC of CD19+CD3-/Day7: number analyzed (Participants) | 14 | 27
  AC of CD19+CD3-/Day7 | 0.31 (0.20) | 0.33 (0.18)
  AC of CD3+CD119+/Day1 | 1.39 (0.67) | 1.53 (1.09)
  AC of CD3+CD119+/Day3: number analyzed (Participants) | 19 | 30
  AC of CD3+CD119+/Day3 | 1.98 (0.7) | 1.85 (0.58)
  AC of CD3+CD119+/Day7: number analyzed (Participants) | 14 | 25
  AC of CD3+CD119+/Day7 | 2.37 (0.94) | 2.39 (0.62)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (leukocytes); Test type: Superiority; p = 0.364, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (leukocytes); Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day1 to day 3 (neutrophils); Test type: Superiority; p = 0.607, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (neutrophils); Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (lymphocytes); Test type: Superiority; p = 0.759, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (lymphocytes); Test type: Superiority; p = 0.777, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (monocytes); Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (lymphocytes); Test type: Superiority; p = 0.343, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (eosinophils); Test type: Superiority; p = 0.575, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (eosinophils); Test type: Superiority; p = 0.912, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (basophils); Test type: Superiority; p = 0.242, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (basophils); Test type: Superiority; p = 0.102, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD3+); Test type: Superiority; p = 0.429, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD3+); Test type: Superiority; p = 0.783, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD3+CD4+); Test type: Superiority; p = 0.466, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD3+CD4+); Test type: Superiority; p = 0.945, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD3+CD8+); Test type: Superiority; p = 0.335, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD3+CD8+); Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD3+CD16+CD56+); Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD3+CD16+CD56+); Test type: Superiority; p = 0.573, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD3-CD16+CD56+); Test type: Superiority; p = 0.472, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD3-CD16+CD56+); Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD3-CD8+); Test type: Superiority; p = 0.727, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD3-CD8+); Test type: Superiority; p = 0.554, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD19+CD3-); Test type: Superiority; p = 0.837, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD19+CD3-); Test type: Superiority; p = 0.967, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (CD3+CD119+); Test type: Superiority; p = 0.473, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (CD3+CD119+); Test type: Superiority; p = 0.736, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Dynamics of Parameters of Immune Status (Relative Percentage of Each Type of White Blood Cells and Different Lymphocyte Phenotypes).
Description: The relative percentage of each type of white blood cells (WBC): Relative Count (AC) of leukocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils, and CD3, CD4, CD8, CD4/CD8, CD16, CD119 leukocytes.
Time Frame: On days 1, 3 and 7 of observation.
Population: Intention to treat [ITT]
Measure: Mean (Standard Deviation); unit: Percentage of total white blood cells
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
Number analyzed (Participants) | 19 | 31
Percentage of total white blood cells
  RC of neutrophils/Day1: number analyzed (Participants) | 18 | 27
  RC of neutrophils/Day1 | 60.59 (12.71) | 55.60 (11.82)
  RC of neutrophils/Day3: number analyzed (Participants) | 15 | 27
  RC of neutrophils/Day3 | 47.59 (9.03) | 45.83 (11.09)
  RC of neutrophils/Day7: number analyzed (Participants) | 15 | 22
  RC of neutrophils/Day7 | 47.94 (11.48) | 52.53 (11.05)
  RC of lymphocytes/Day1: number analyzed (Participants) | 19 | 29
  RC of lymphocytes/Day1 | 25.97 (11.78) | 24.42 (10.03)
  RC of lymphocytes/Day3: number analyzed (Participants) | 18 | 31
  RC of lymphocytes/Day3 | 40.72 (8.10) | 41.99 (12.26)
  RC of lymphocytes/Day7: number analyzed (Participants) | 18 | 27
  RC of lymphocytes/Day7 | 42.95 (10.87) | 38.69 (10.09)
  RC of monocytes/Day1: number analyzed (Participants) | 19 | 29
  RC of monocytes/Day1 | 11.53 (5.01) | 13.97 (4.04)
  RC of monocytes/Day3: number analyzed (Participants) | 18 | 31
  RC of monocytes/Day3 | 11.76 (3.76) | 10.92 (3.58)
  RC of monocytes/Day7: number analyzed (Participants) | 18 | 27
  RC of monocytes/Day7 | 8.36 (2.56) | 7.64 (2.00)
  RC of eosinophils/Day1: number analyzed (Participants) | 19 | 29
  RC of eosinophils/Day1 | 1.05 (1.07) | 1.32 (1.55)
  RC of eosinophils/Day3: number analyzed (Participants) | 18 | 31
  RC of eosinophils/Day3 | 1.28 (1.11) | 2.07 (2.04)
  RC of eosinophils/Day7: number analyzed (Participants) | 18 | 27
  RC of eosinophils/Day7 | 1.86 (1.53) | 1.85 (1.65)
  RC of basophils/Day1: number analyzed (Participants) | 19 | 29
  RC of basophils/Day1 | 0.48 (0.30) | 0.76 (0.56)
  RC of basophils/Day3: number analyzed (Participants) | 18 | 31
  RC of basophils/Day3 | 0.46 (0.32) | 0.58 (0.40)
  RC of basophils/Day7: number analyzed (Participants) | 18 | 27
  RC of basophils/Day7 | 0.61 (0.42) | 0.41 (0.29)
  RC of CD3+/Day1 | 74.08 (15.28) | 75.69 (8.14)
  RC of CD3+/Day3: number analyzed (Participants) | 19 | 30
  RC of CD3+/Day3 | 80.62 (7.26) | 79.75 (7.82)
  RC of CD3+/Day7: number analyzed (Participants) | 14 | 28
  RC of CD3+/Day7 | 80.07 (10.04) | 78.44 (9.15)
  RC of CD3+CD4+/Day1 | 46.63 (13.95) | 48.32 (9.83)
  RC of CD3+CD4+/Day3: number analyzed (Participants) | 19 | 30
  RC of CD3+CD4+/Day3 | 51.87 (7.87) | 51.33 (9.29)
  RC of CD3+CD4+/Day7: number analyzed (Participants) | 14 | 28
  RC of CD3+CD4+/Day7 | 52.06 (10.16) | 51.55 (11.63)
  RC of CD3+CD8+/Day1 | 25.80 (11.74) | 23.92 (8.51)
  RC of CD3+CD8+/Day3: number analyzed (Participants) | 19 | 30
  RC of CD3+CD8+/Day3 | 26.36 (8.07) | 25.21 (5.64)
  RC of CD3+CD8+/Day7: number analyzed (Participants) | 14 | 28
  RC of CD3+CD8+/Day7 | 26.49 (7.23) | 24.70 (5.36)
  RC of CD3+CD16+CD56+/Day1 | 4.99 (3.36) | 4.66 (3.48)
  RC of CD3+CD16+CD56+/Day3: number analyzed (Participants) | 19 | 30
  RC of CD3+CD16+CD56+/Day3 | 5.44 (3.18) | 3.78 (2.10)
  RC of CD3+CD16+CD56+/Day7: number analyzed (Participants) | 14 | 28
  RC of CD3+CD16+CD56+/Day7 | 4.24 (3.26) | 3.24 (2.29)
  RC of CD3-CD16+56+/Day1 | 12.33 (10.82) | 9.20 (6.04)
  RC of CD3-CD16+56+/Day3: number analyzed (Participants) | 19 | 30
  RC of CD3-CD16+56+/Day3 | 9.68 (6.29) | 8.88 (6.58)
  RC of CD3-CD16+56+/Day7: number analyzed (Participants) | 14 | 28
  RC of CD3-CD16+56+/Day7 | 7.15 (5.35) | 7.35 (5.27)
  RC of CD3-CD8+/Day1 | 4.38 (4.01) | 3.48 (3.01)
  RC of CD3-CD8+/Day3: number analyzed (Participants) | 19 | 30
  RC of CD3-CD8+/Day3 | 4.06 (2.86) | 3.73 (2.50)
  RC of CD3-CD8+/Day7: number analyzed (Participants) | 14 | 28
  RC of CD3-CD8+/Day7 | 3.55 (2.32) | 3.18 (2.02)
  RC of CD19+CD3-/Day1 | 13.70 (8.70) | 14.96 (7.93)
  RC of CD19+CD3-/Day3: number analyzed (Participants) | 19 | 30
  RC of CD19+CD3-/Day3 | 9.71 (4.05) | 10.79 (4.85)
  RC of CD19+CD3-/Day7: number analyzed (Participants) | 14 | 28
  RC of CD19+CD3-/Day7 | 12.82 (5.45) | 14.56 (7.35)
Statistical Analysis 1: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of neutrophils); Test type: Superiority; p = 0.282, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of neutrophils); Test type: Superiority; p = 0.071, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of lymphocytes); Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of lymphocytes); Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of monocytes); Test type: Superiority; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of monocytes); Test type: Superiority; p = 0.019, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of eosinophils); Test type: Superiority; p = 0.424, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of eosinophils); Test type: Superiority; p = 0.666, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of basophils); Test type: Superiority; p = 0.268, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of basophils); Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of CD3+); Test type: Superiority; p = 0.361, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of CD3+); Test type: Superiority; p = 0.699, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of CD3+CD4+); Test type: Superiority; p = 0.418, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of CD3+CD4+); Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of CD3+CD8+); Test type: Superiority; p = 0.172, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of CD3+CD8+); Test type: Superiority; p = 0.904, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of CD3+CD16+CD56+); Test type: Superiority; p = 0.148, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of CD3+CD16+CD56+); Test type: Superiority; p = 0.821, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of CD3-CD16+CD56+); Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of CD3-CD16+CD56+); Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of CD3-CD8+); Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of CD3-CD8+); Test type: Superiority; p = 0.821, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 3 (RC of CD19+CD3-); Test type: Superiority; p = 0.943, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Ergoferon (1 Tablet 3 Times a Day) vs Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day; difference between changes from day 1 to day 7 (RC of CD19+CD3-); Test type: Superiority; p = 0.841, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were collected for 7 days (5 days of the therapy plus follow-up period).
Description: Adverse/Serious adverse events were collected in patients of the Safety population (n=184)
Arm/Group | Ergoferon (1 Tablet 3 Times a Day) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/92
Other Adverse Events (participants affected / at risk) | 10/92 | 10/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ergoferon (1 Tablet 3 Times a Day) (N=92) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day (N=92)
Hyperthermia (General disorders) | 1 | 0 — Hyperthermia was recorded as a serious adverse event (SAE) because the patient was hospitalized. The outcome of SAE is recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ergoferon (1 Tablet 3 Times a Day) (N=92) | Oseltamivir (Tamiflu) - 1 Capsule (75mg) Two Times a Day (N=92)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 2
Lacrimation increased (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Chest pain (General disorders) | 1 | 1
Hyperthermia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT01850446/Prot_SAP_000.pdf